CLINICAL TRIAL: NCT00638586
Title: Comparison of Patients Undergoing Radial or Femoral Arterial Access for Percutaneous Catheterization-Nursing Aspects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: HY/102008
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Femoral Artery Access; Radial Artery Access

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Femoral access
- 2: Radial access

SUMMARY:
Transradial access is a recently developed alternative for diagnostic andf interventional cardiac catheterization. We sought to compare the differences between patients that have undergone PTCA transradial and transfemoral access from the nursing point of view:

1. Anxiety levels
2. Pain at access point, pain in general and level of pain during mobility
3. Differences in feelings of embarrassement
4. Differences in satisfaction

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for PTCA without any exclusion criteria

Exclusion Criteria:

* Dementia
* Psychiatric patients
* Unconscious
* Minors
* Patients who had PTCA in past
* Patients who were initially scheduled for different access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hospitalized patients that are candidates for undergoing PTCA.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2008-04

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel